CLINICAL TRIAL: NCT03142360
Title: Effect of Beraprost Sodium (Berasil) on Hemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2017-0129
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Arteriovenous Fistula Patency
MeSH Terms: interventions — beraprost

STUDY DESIGN:
Intervention Model Description: Treatment group is randomly assigned to start taking 120 mcg of Berasil. On the other hand, the control group does not take anything.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Within two days after successful arteriovenous graft surgery, the treatment group is randomly assigned to start taking 120 mcg of Berasil.
  Interventions: Drug: Beraprost sodium (Berasil)
- Non-Treatment group (No Intervention): On the other hand, the control group does not take anything.

INTERVENTIONS:
Drug: Beraprost sodium (Berasil) — Within two days after successful arteriovenous graft surgery, the treatment group is randomly assigned to start taking 120 mcg of Berasil.
  Arms: Treatment group

SUMMARY:
There is no randomized control study to determine if the beneficial effects of beraprost sodium could improve the patency of arteriovenous fistula in hemodialysis patients. Therefore, this study is aimed to demonstrate the use of beraprost sodium can improve the patency of arteriovenous fistula in patients undergoing hemodialysis. This study is prospectively randomize controlled open-label trials in patients who newly made artificial arteriovenous fistula for hemodialysis. This study is a pilot study, and the target number of subjects is 60 in total, 30 in the treatment group and 30 in the control group.

After randomization, the treatment group takes a beraprost sodium for 6 months and the control group does not take placebo.

Treatment lasts for 6 months after dosing but continues until the patient changes the renal-replacement therapy method or falls under the exclusion criteria.

The patient should visit at 1, 3, and 6 months after arteriovenous graft surgery to check the access site after graft surgery. The doppler ultrasound test is performed to measure the access blood flow rate and patency of arteriovenous fistula.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled open-labeled trial of patients undergoing hemodialysis under the diagnosis of end stage renal disease. The subjects were divided into the treatment group and the control group through random assignment under the condition of receiving hemodialysis steadily and followed up for 6 months. After randomization, the treatment group received beraprost sodium (Berasil) for 6 months (24 weeks) and beraprost sodium will be provided by Astellas Pharma Korea, Inc. Patients were randomly assigned within 2 days after successful arteriovenous graft surgery, and the treatment group started taking 120 mcg of Berasil, while the control group did not take placebo to replace beraprost sodium.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet all of the following criteria

  1. Patient who newly made artificial arteriovenous fistula for hemodialysis
  2. Patients who agree to participate in the test and sign a consent form
  3. Patients who had diabetes

Exclusion Criteria:

* Patients under 18 years old, 80 years old or older
* Patients with a high risk of bleeding (hemophilia, capillary weakness, upper gastrointestinal bleeding, urinary tract bleeding, hemoptysis, vitreous hemorrhage, etc.)
* Women who are pregnant or have a possibility of pregnancy
* Platelet count ≤ 75000
* Patients taking anticoagulants or antithrombotics
* Patients with galactose intolerance, lactase deficiency or glucose-galactose malabsorption

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-04-05 (Actual); Primary Completion 2019-04-04 (Estimated); Study Completion 2019-04-04 (Estimated)

PRIMARY OUTCOMES:
AVF maturation rate | 3 months after arteriovenous graft surgery
  Physiologic maturation of the AVF by the definition of AVF access blood flow ≥500mlL/min and AVF diameter ≥4mm at 3 months

SECONDARY OUTCOMES:
AVF maturation rate | 1 month after arteriovenous graft surgery
  Physiologic maturation of the AVF by the definition of AVF access blood flow ≥500mlL/min and AVF diameter ≥4mm at a month
Hemodialysis performed rate | 3 months after arteriovenous graft surgery
AVF failure rate | 6 months after arteriovenous graft surgery
Bleeding events | 6 months after arteriovenous graft surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Nephrology, Department of Internal Medicine Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin CC, Yang WC, Chen MC, Liu WS, Yang CY, Lee PC. Effect of far infrared therapy on arteriovenous fistula maturation: an open-label randomized controlled trial. Am J Kidney Dis. 2013 Aug;62(2):304-11. doi: 10.1053/j.ajkd.2013.01.015. Epub 2013 Mar 6. PMID 23474008
- [Background] Na KY, Kim DK, Kim SG, Lee YK, Lim CS. Effect of beraprost sodium on arterial stiffness in patients with type 2 diabetic nephropathy. Trials. 2013 Sep 2;14:275. doi: 10.1186/1745-6215-14-275. PMID 24066672
- [Background] Dixon BS, Beck GJ, Vazquez MA, Greenberg A, Delmez JA, Allon M, Dember LM, Himmelfarb J, Gassman JJ, Greene T, Radeva MK, Davidson IJ, Ikizler TA, Braden GL, Fenves AZ, Kaufman JS, Cotton JR Jr, Martin KJ, McNeil JW, Rahman A, Lawson JH, Whiting JF, Hu B, Meyers CM, Kusek JW, Feldman HI; DAC Study Group. Effect of dipyridamole plus aspirin on hemodialysis graft patency. N Engl J Med. 2009 May 21;360(21):2191-201. doi: 10.1056/NEJMoa0805840. PMID 19458364
- [Background] Vicil S, Erdogan S. Beraprost sodium, a prostacyclin (PGI) analogue, ameliorates lipopolysaccharide-induced cellular injury in lung alveolar epithelial cells. Turk J Med Sci. 2015;45(2):284-90. doi: 10.3906/sag-1401-108. PMID 26084116
- [Background] Arai T. Long-term effects of beraprost sodium on arteriosclerosis obliterans: a single-center retrospective study of Japanese patients. Adv Ther. 2013 May;30(5):528-40. doi: 10.1007/s12325-013-0030-7. Epub 2013 Jun 8. PMID 23749750
- [Background] Murakami M, Watanabe M, Furukawa H, Nakahara H. The prostacyclin analogue beraprost sodium prevents occlusion of bypass grafts in patients with lower extremity arterial occlusive disease: a 20-year retrospective study. Ann Vasc Surg. 2005 Nov;19(6):838-42. doi: 10.1007/s10016-005-7668-9. PMID 16247707
- [Background] Sakao S, Tanabe N, Kasahara Y, Tatsumi K. Long-term survival of Japanese patients with pulmonary arterial hypertension treated with beraprost sodium, an oral prostacyclin analogue. Intern Med. 2014;53(17):1913-20. doi: 10.2169/internalmedicine.53.2573. Epub 2014 Sep 1. PMID 25175122